CLINICAL TRIAL: NCT04106895
Title: Use of Fibryga, a Fibrinogen Concentrate in Real World: Retrospective Collection of Clinical Data
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: FORMA-10
Record Dates: First submitted 2019-08-28; First posted 2019-09-27 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fibryga
  Interventions: Drug: Fibryga

INTERVENTIONS:
Drug: Fibryga — Fibryga

SUMMARY:
To describe the characteristics of patients treated with Fibryga®, the indications and conditions of use of Fibryga® and, for patients treated " on-demand", the short-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with fibrinogen deficiency (congenital or acquired)
* Having received an treatment with Fibryga® during the recollection period
* Having been informed of the potential retrospective collection of their data by a Clinical Research Associate mandated by Octapharma® when Fibryga® has been delivered and who did not refuse.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having received Fibryga® ("on-demand" or for regular prophylaxis) in the centres participating in the study during the recollection period (limited to 7 patients by centre and by period). A total of 4 recollection periods is planned by centre.
  Data from all consecutive patients having received Fibryga® whatever the indication (congenital or acquired fibrinogen deficiency; "on-demand" or regular prophylaxis) will be collected. The data collection will be limited to 7 patients by centre and by period, meaning that only data from the 7 first patients treated during the recollection period willbe collected.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
proportion of treatments given for an ongoing bleeding episodes | 6 months
  Estimate the proportion of treatments given for an ongoing bleeding episodes (opposed to preventative treatment administered for example before surgery or to regular prophylaxis)

SECONDARY OUTCOMES:
On-demand Treatment Success | 6 months
  on-demand treatment of spontaneous or surgical bleeding episodes, success is defined as bleeding control (complete cessation of bleeding or < 20% decrease in hemoglobin).
Surgical Prophylaxis Success | 6 months
  Surgical prophylaxis success is defined as no bleeding or oozing and control of bleeding with fibrinogen concentrate (as anticipated or requiring increased dosing or additional infusions not originally anticipated).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Bordeaux Study Site, Bordeaux
  - Le Plessis Robinsin Study Site, Le Plessis-Robinson
  - Marseille Study Site, Marseille
  - Nantes Study Site, Nantes
  - Valence Study Site, Valence

IPD SHARING:
Plan to Share IPD: Undecided